CLINICAL TRIAL: NCT01662947
Title: Verify Wrist BPM TMB-1117 to Comply With ANSI/AAMI SP10
Brief Title: Clinical Study of Wrist Blood Pressure Monitor in Conformance With the ANSI/AAMI SP10 Standard
Acronym: WristBPM01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leo Wang (Other)
Collaborators: BTS International (Other)
Responsible Party: Sponsor-Investigator, Leo Wang, Team leader, BTS International
Organization: BTS International (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: Wrist BPM TMB-1117; BTS-TRANS12001 (Other: BTSInternational)
Record Dates: First submitted 2012-08-01; First posted 2012-08-13 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Efficacy of Wrist BPM Measurement; Hypertension
Keywords: blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DUT Arm (Experimental): DUT: Transtek Wrist Blood Pressure Monitor TMB-1117
  Measurement: Blood Pressure
  Groups/Cohorts: DUT
  Interventions: Device: Blood pressure Transtek Wrist Blood Pressure Monitor, TMB-1117
- Reference Arm (Experimental): Reference Device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1mmHg and range: 0-300mmHg.
  Measurement: Blood Pressure
  Groups/Cohorts: Reference
  Interventions: Device: Blood pressure Reference Device: Yuyue Medical Blood Pressure Meter, YYBP-2

INTERVENTIONS:
Device: Blood pressure Transtek Wrist Blood Pressure Monitor, TMB-1117 — Systolic, Diastolic pressure.
  Other Names: DUT TMB-1117 measurement
  Arms: DUT Arm
Device: Blood pressure Reference Device: Yuyue Medical Blood Pressure Meter, YYBP-2 — Systolic, Diastolic pressure
  Other Names: Reference mercury sphygmomanometer measurement
  Arms: Reference Arm

SUMMARY:
The clinical protocol of the clinical testing of this device:

1. Objective of the test: To verify the efficiency of device.
2. Test methods and procedures: Clinical test in two positions: Seated and Supine.
3. DUT: Transtek Wrist Blood Pressure Monitor, Model: TMB-1117. Cuff size: 13.5 - 21.5 cm.
4. Comparison device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1 mmHg and range: 0-300 mmHg.
5. Study endpoints: Comply with ANSI/AAMI SP10-2002 standard.
6. Statistical methodology used: Description of statistical methods.
7. Result: Meet the requirements of SP10.

DETAILED DESCRIPTION:
Hospital Information

Hospital Information The data was collected by Zhongshan City People's Hospital Clinical Investigator Team at Zhongshan City People's Hospital, No.2 Sunwen Dong Road, Zhongshan, Guangdong 528403, P. R. China.

Investigator: Dr. Cao Yuedong, Leader; Li Qidong, Nurse A; Chen Wenqian, Nurse B.

Contact Dr. Cao Yuedong Tel: +86 760 88823818

Used Equipments DUT (Device Under Test): Transtek Wrist Blood Pressure Monitor, TMB-1117 Reference Device: Yuyue Medical Blood Pressure Meter, YYBP-212, accuracy: ±1 mmHg and range: 0-300 mmHg.

Test Protocol

1. Test Purpose:

   The aim of clinical test is to determine, for the purpose of design qualification, the overall performance of the system meeting the following requirement: For systolic and diastolic pressures, treated separately, the mean difference of the paired measurement of the test system and the comparison system shall be ± 5 mmHg or less, with standard deviation of 8 mmHg or less.
2. Target Subject:

1) The subject database shall contain at least 85 subjects. 2) The distribution of blood pressure of the subjects required to be: At least 10 percent below 100 mmHg systolic; at least 10 percent above 160 mmHg systolic; at least 10 percent below 60 mmHg diastolic; at least 10 percent above 100 mmHg diastolic; with the remainder distributed between these outer limits.

3. Identification and precision of equipment used According to ANSI/AAMI SP10, the maximum measurement error of the non-automatic sphygmomanometers used in the comparing test shall not exceed 1.0mmHg at the temperature of the test. The manometer was used to verify its accuracy before test.

The clinical study was conducted according to the protocol described in the ANSI/AAMI SP10 with 85 subjects.

4. Test procedures (auscultatory method, same-limb sequential measurement was chosen)

1. Record the age, gender, and circumference of the left wrist of the subject.
2. Let subject seated or supine calmly for five minutes before test.
3. Measure heart rate in one minute by palpation on radial artery, record it.
4. Two observers shall make simultaneous, blinded, blood pressure determination on the subject's left arm. Each nurse will write down the reading on a small piece of paper, make a tick if there is an auscultatory gap and then submit to the recorder.
5. The two readings separately from two observers will be recorded, and if two observers agree that they find an auscultatory gap this time, it will also be recorded. The wrist cuff will be take off, after 90 seconds rest, TMB-1117 cuff will be taken on and tested, and the readings (systolic, diastolic, mean BP and Heart rate) be recorded.
6. For each subject, repeat 3) and 5) to get 3 measurements.
7. Repeat step 1) to 6) for every subject.

5. Note:

1. No motion and speaking are allowed during the measurement.
2. The reference device's cuff release at the rate about 3 mmHg/s so to ensure an accurate reading of observer.
3. The arm, wrist and the haear of subject to keep on the same height when measurement.
4. Test environment: Temperature: 20±1 ℃; Relative humidity: 40~50%.

ELIGIBILITY:
Inclusion Criteria:

* male,female,

Exclusion Criteria:

* below 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Verify the accuracy of measure functions of device | 10 days
  Verify the accuracy of device if meet the requirements of ANSI/AAMI SP10 when it measure Systolic & Diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Leo Wang, Leader, Study Chair — BTS International
Locations (1):
- Zhongshan City People's Hospital, Zhongshan, Guangdong, China

REFERENCES:
- [Background] Alpert BS. Validation of the Tiba Medical Ambulo 2400 ambulatory blood pressure monitor to the ISO Standard and BHS protocol. Blood Press Monit. 2010 Oct;15(5):275-7. doi: 10.1097/MBP.0b013e32833c8b39. PMID 20559140
- See also: Related Info — http://www.zsph.com